CLINICAL TRIAL: NCT06513156
Title: Continuum of Care in Hospitalized Patients With Opioid or Stimulant Use Disorder and Infectious Complications of Drug Use - Substance Use/ID Integrated Clinic vs. TAU to Prevent Infection Related Readmission
Brief Title: Continuum of Care in Hospitalized Patients With Opioid/Stimulant Use Disorder and Infectious Complications From Drug Use
Acronym: CHOICE-STAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Elana Rosenthal (Other)
Collaborators: Emory University (Other); George Washington University (Other); West Virginia University (Other); Weill Medical College of Cornell University (Other); Friends Research Institute, Inc. (Other)
Responsible Party: Sponsor-Investigator, Elana Rosenthal, Associate Professor, University of Maryland, Baltimore
Organization: University of Maryland, Baltimore (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00111318
Record Dates: First submitted 2024-07-08; First posted 2024-07-22 (Actual); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder; Injection Related Infections; Stimulant Use Disorder
Keywords: Delivery of Health Care, Integrated; Opioid use disorder; Serious Injection Related Infections; Stimulant Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment As Usual (No Intervention): Will receive treatment for infection and opioid or stimulant use disorder per the usual care at each hospital
- Integrated Infectious Diseases and Substance Use Disorder Clinic (IC) (Experimental): The Integrated ID/SUD Clinic will provide facilitated linkage to a clinic providing medical treatment aimed at treating SUD, resolving the sentinel infection, treating existing ID complications of OUD/stimulants (HIV, HCV, wounds) and preventing subsequent infections by providing accessible care for infectious diseases and MOUD treatment that is integrated into a single appointment and co-located at a single site (either in person or via telemedicine) for a minimum of monthly appointments over a 6 month time period. A feature of the IC will be weekly care coordination meetings between the ID and SUD providers. The dual goals of the IC intervention are to 1) to facilitate accessibility to ID and OUD care and 2) to ensure care coordination between outpatient ID and SUD providers.
  Interventions: Behavioral: Integrated Infectious Diseases and Substance Use Disorder Clinic (IC)

INTERVENTIONS:
Behavioral: Integrated Infectious Diseases and Substance Use Disorder Clinic (IC) — Integrated medication for opioid/stimulant use disorder and infectious disease care provided into single appointment either in person or via telemedicine with a minimum of monthly appointments for 6 months.
  Arms: Integrated Infectious Diseases and Substance Use Disorder Clinic (IC)

SUMMARY:
This is a two-group randomized controlled trial conducted at five hospitals across the U.S. designed to test the effectiveness of an Integrated infectious diseases/Substance Use Disorder outpatient clinic (IC) compared to treatment as usual aimed at reducing infection related readmissions and improving health outcomes in people hospitalized with an infection related to injecting opioids or stimulants.

DETAILED DESCRIPTION:
This is a phase III two arm randomized controlled trial to determine the impact and Integrated infectious diseases (ID) and Substance Use Disorder outpatient clinic (IC) compared to treatment as usual on infection related rehospitalization in individuals hospitalized with infections due to injecting opioids or Stimulants, in the 6 month time period after discharge. This study includes both cost effectiveness and implementation outcomes.

(1) IC will provide facilitated linkage to a clinic providing medical treatment aimed at treating substance use disorder (SUD), resolving the index infection, treating existing ID complications of OUD (HIV, HCV, wounds) and preventing subsequent infections by providing accessible care for infectious diseases and medication for OUD (MOUD) treatment that is integrated into a single appointment and co-located at a single site (either in person or via telemedicine) for a minimum of monthly appointments over a 6 month time period. A feature of the IC will be weekly care coordination meetings between the ID and MOUD providers.

The study will recruit patients during hospitalization for an infection due to injecting opioids or stimulants at four hospital systems (five hospitals) and randomly assign approximately 304 inpatients in 1:1 ratio to IC vs TAU.

Participants will be followed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Admitted to study hospital (defined as hospitalized with a primary team that is not Emergency Medicine)
3. Injection opioid or stimulant use in past 90 days - per patient self-report
4. Active suspected or confirmed qualifying infection (see list) at time of admission.

Qualifying infections:

* Non-vertebral osteomyelitis
* Vertebral osteomyelitis or discitis
* Epidural, subdural, or extradural abscess
* Intracranial or intraspinal abscess
* Native joint septic arthritis
* Prosthetic joint septic arthritis
* Blood stream infection (bacterial or fungal)
* Native valve Endocarditis
* Prosthetic valve endocarditis
* Cardiac Implantable electronic device infection
* Infectious pseudoaneurysm and aneurysm
* Infected vascular graft
* Septic venous thrombosis
* Skin and Soft tissue infection (cellulitis, skin abscess, necrotizing fasciitis)
* Infected skin ulcer
* Orthopedic hardware infection
* Muscle abscess/myositis
* Central nervous system infection (bacterial or fungal)
* Bacterial or fungal ophthalmologic infection
* Other abscess
* Pulmonary septic emboli
* Other acute bacterial or fungal infection deemed appropriate by site study team

Exclusion Criteria:

* 1. Infection due to a cause other than injection drug use, per determination of a site PI.

  2. Inability to provide consent due to circumstance (e.g., sedated, intubated), language, or cognitive impairment.

  3. Unwilling to provide informed consent 4. Unable to receive potential interventions due to geography 5. On comfort measures or planned for discharge to hospice care 6. Incarcerated at the time of hospitalization 7. Other criteria at the discretion of the site investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 304 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2027-07-30 (Estimated)

PRIMARY OUTCOMES:
Infection Rehospitalization | 6 months after discharge for index hospitalization
  New hospitalization due to infection following discharge for index hospitalization

SECONDARY OUTCOMES:
Time to first infection related readmission | 12 months after discharge for index hospitalization
  Time to first infection related readmission
Reason for infection related readmission | 12 months after discharge for index hospitalization
  Reason for infection related readmission (persistent index infection, new IDU associated infection, other infection)
Hospital services utilization | 12 months after discharge for index hospitalization
  ED visits (Binary, count, time to first ED visit, cause) and Readmission, all cause (binary, count, time to first readmission, cause)
Mortality | 12 months after discharge for index hospitalization
  Death (Binary, time to death, cause of death)
Index infection | 3 months after discharge for index hospitalization
  Completion of antibiotics (binary, reason for incomplete antibiotics); Resolution of index infection (binary) Skilled Nursing Facility (SNF) Admitted to SNF (binary) Discharge type from SNF (planned, PDD, dead, transfer)
Other Infections | 12 months after discharge for index hospitalization
  HCV Active HCV (binary) Clinical evaluation (binary) DAA prescribed (binary) DAA initiated (binary) SVR achieved (binary) HIV Diagnosis status (binary) HIV VL undetectable (binary) ART Taking (binary) Type (pills vs injections) Adherence (# missed doses in last 30 days) PrEP Eligible (CDC Criteria, binary, indication) Offered by healthcare provider (binary) Taking (binary) Type (pills vs injections) Adherence (# missed doses in last 30 days)
Skin and soft tissue wounds | 12 months after discharge for index hospitalization
  Present (binary) Number (count) Per wound Size Location on body Duration (continuous)
New infections not requiring hospitalization | 12 months after discharge for index hospitalization
  * Present (binary)
  * Number (count)
Outpatient linkage and retention | 12 months after discharge for index hospitalization
  * Infectious Diseases Clinic (binary, time to linkage, count)
  * Medication for OUD Treatment (binary, time to linkage, count)
  * Non-medication based OUD Treatment (binary, time to linkage, count)
Medication for Opioid Use (MOUD) | 12 months after discharge for index hospitalization
  * On treatment (binary)
  * MOUD type
  * MOUD Dose
  * MOUD Dose adequacy
  * MOUD Source of medication
  * MOUD Location type
  * MOUD Co-location with other services
  * Reasons for no MOUD (descriptive)
Medication for stimulant use (MStUD) | 12 months after discharge for index hospitalization
  * On treatment (binary) MStUD type
  * MStUD Dose
  * MStUD Dose adequacy
  * MStUD Source of medication
  * MStUD Location type
  * MStUD Co-location with other services
  * Reasons for no MStUD (descriptive)
Substance Use-Opioid | 12 months after discharge for index hospitalization
  Ongoing opioid (binary, mode)
  * Opioid use frequency
  * Mode of opioid use
  * Opioid craving
  * Other drug use (binary, mode)
  * Other drug use frequency
  * IDU (binary, frequency, mode (IM, IV, skin, other), location, syringe reuse, ssp engagement).
  * Severity (DAST)
  * Overdose (binary, count)
  * Tobacco use
  * UDS (binary - presence of opioids, )
Substance Use - Stimulant | 12 months after discharge for index hospitalization
  Ongoing stimulant use (binary, mode)
  * Stimulant use frequency
  * Mode of stimulant use
  * Cocaine craving
  * Methamphetamine craving
  * Other drug use (binary, mode)
  * Other drug use frequency
  * IDU (binary, frequency, mode (IM, IV, skin, other), location, syringe reuse, ssp engagement).
  * Severity (DAST)
  * Overdose (binary, count)
  * Tobacco use
  * UDS (binary - presence of cocaine, amphetamines, other)
Cost Effectiveness | 12 months after discharge for index hospitalization
  • ICER for quality adjusted life years (QALYs); opioid-free years (OfYs); and infection-free years (IfYs) gained

CONTACTS AND LOCATIONS:
Overall Officials: Elana Rosenthal, MD, Principal Investigator — University of Maryland, Baltimore
Locations (4):
- United States (4):
  - George Washington University, Washington D.C., District of Columbia
  - Emory University, Atlanta, Georgia
  - University of Maryland Baltimore, Baltimore, Maryland
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No